CLINICAL TRIAL: NCT01101763
Title: A Pilot Study to Evaluate the Plasma Enrichment Kinetics of a 13C-Cholesterol Infusate in Healthy Male Subjects
Brief Title: A Study of the Kinetics of a 13C-Cholesterol Infusate in Healthy Male Subjects (0000-108)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-108; 108; 2010_022
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Subjects: Healthy males

SUMMARY:
This is a 2-part pilot study in healthy male subjects to evaluate plasma enrichment kinetics of [13C3,4]-cholesterol (Part I) and to assess the test-retest reproducibility (Part II) of Reverse Cholesterol Transport (RCT) measurements. The study will determine whether atom percent enrichment (% APE) at 18 hours can be extrapolated from the steady-state value and whether the mean difference in repeat Ra measurements is below is a prespecified level.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male 18 to 45 years of age at screening
* Subject has a stable weight (± 2 kg) for more then 6 weeks prior to screening

Exclusion Criteria:

* Subject has a history of ileal bypass, gastric bypass, or other significant condition associated with malabsorption
* Subject has an active or recent (<2 weeks) gastrointestinal condition (gastroenteritis, diarrhea, chronic constipation, irritable bowl syndrome, etc.) affecting bowel movements
* Subject has a known allergy to beans, peas, eggs or egg-derived products and/or soy or soy-derived products
* Subject has a history of plant sterol storage disease (sitosterolemia, cerebrotendinotic xanthomatosis) or a history of intolerance to plant sterols and/or plant sterol containing products
* Subject has a history of hepatic or gall bladder disease (including gallstones, cholecystectomy, etc.)
* Subject is currently taking psyllium, other fiber-based laxatives, phytosterol margarines, and/or over the counter (OTC) therapies that are known to affect serum lipids
* Subject has taken lipid-lowering agents within 6 weeks prior to screening
* Subject has previously been administered an intravenous infusion of [13C3,4]-cholesterol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited for the study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
%APE (atom percent enrichment) for all study subjects in Part I at 18 hours | 18 hours
Rate of appearance (Ra) of unlabeled cholesterol from the whole-body peripheral pool | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC